CLINICAL TRIAL: NCT00751881
Title: A Multi-center Double-blind Parallel-group Placebo-controlled Study of the Efficacy and Safety of Teriflunomide in Patients With Relapsing Multiple Sclerosis
Brief Title: An Efficacy Study of Teriflunomide in Participants With Relapsing Multiple Sclerosis
Acronym: TOWER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC10531; 2007-004452-36 (EudraCT Number)
Record Dates: First submitted 2008-05-07; First posted 2008-09-12 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis
Keywords: relapsing multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Teriflunomide 7 mg / 14 mg (Experimental): Core treatment period: Teriflunomide 7 mg once daily. Extension treatment period: Teriflunomide 14 mg once daily.
  Interventions: Drug: Teriflunomide
- Teriflunomide 14 mg / 14 mg (Experimental): Core treatment period: Teriflunomide 14 mg once daily. Extension treatment period: Teriflunomide 14 mg once daily.
  Interventions: Drug: Teriflunomide
- Placebo / Teriflunomide 14 mg (Placebo Comparator): Core treatment period: Placebo (for teriflunomide) once daily. Extension treatment period: Teriflunomide 14 mg once daily.
  Interventions: Drug: Placebo; Drug: Teriflunomide

INTERVENTIONS:
Drug: Placebo — Film-coated tablet
  Oral administration
  Arms: Placebo / Teriflunomide 14 mg
Drug: Teriflunomide — Film-coated tablet
  Oral administration
  Other Names: HMR1726

SUMMARY:
The primary objective of the study was to assess the effect of two doses of teriflunomide, in comparison to placebo, on the frequency of multiple sclerosis (MS) relapses in participants with relapsing MS.

Key secondary objective was to assess the effect of the two doses of teriflunomide, in comparison to placebo, on disability progression.

Other secondary objectives were:

* To assess the effect of the two doses of teriflunomide in comparison to placebo on:

  * Fatigue;
  * Health-related quality of life, a measure of the impact of the participant's health on his or her overall well being.
* To evaluate the safety and tolerability of teriflunomide.

DETAILED DESCRIPTION:
The study consists of:

* A core treatment period: Teriflunomide 7 mg or Teriflunomide 14 mg or placebo was administered in double-blind fashion until a fixed common end date which was approximately 48 weeks after randomization of the last participant.
* An extension treatment period: the highest dose of teriflunomide was administered in open-label fashion to participants who successfully complete the core treatment period and wish to continue.

The overall treatment period was followed by a 4-week elimination follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing multiple sclerosis,
* Two relapses in prior 2 years or one relapse in prior year.

Exclusion Criteria:

* Clinically relevant cardiovascular, hepatic, neurological, endocrine or other major systemic disease,
* Significantly impaired bone marrow function or, significant anemia, leukopenia or thrombocytopenia,
* Pregnant or nursing woman,
* Alcohol or drug abuse,
* Prior or concomitant use of cladribine, mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporin, methotrexate or mycophenolate,
* Human immunodeficiency virus (HIV) positive,
* Any known condition or circumstance that would prevent, in the investigator's opinion, compliance or completion of the study.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1169 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (193):
- United States (39):
  - Sanofi-Aventis Investigational Site Number 840041, Phoenix, Arizona
  - Sanofi-Aventis Investigational Site Number 840084, Tucson, Arizona
  - Sanofi-Aventis Investigational Site Number 840008, Loma Linda, California
  - Sanofi-Aventis Investigational Site Number 840034, Modesto, California
  - Sanofi-Aventis Investigational Site Number 840090, Fort Collins, Colorado
  - Sanofi-Aventis Investigational Site Number 840011, Fairfield, Connecticut
  - Sanofi-Aventis Investigational Site Number 840013, Maitland, Florida
  - Sanofi-Aventis Investigational Site Number 840083, Ocala, Florida
  - Sanofi-Aventis Investigational Site Number 840086, Ormond Beach, Florida
  - Sanofi-Aventis Investigational Site Number 840025, Sarasota, Florida
  - Sanofi-Aventis Investigational Site Number 840015, St. Petersburg, Florida
  - Sanofi-Aventis Investigational Site Number 840033, Sunrise, Florida
  - Sanofi-Aventis Investigational Site Number 840063, Elk Grove Village, Illinois
  - Sanofi-Aventis Investigational Site Number 840064, Flossmoor, Illinois
  - Sanofi-Aventis Investigational Site Number 840039, Fort Wayne, Indiana
  - Sanofi-Aventis Investigational Site Number 840012, Indianapolis, Indiana
  - Sanofi-Aventis Investigational Site Number 840016, Des Moines, Iowa
  - Sanofi-Aventis Investigational Site Number 840069, Clinton Township, Michigan
  - Sanofi-Aventis Investigational Site Number 840075, Grand Rapids, Michigan
  - Sanofi-Aventis Investigational Site Number 840061, Traverse City, Michigan
  - Sanofi-Aventis Investigational Site Number 840076, Minneapolis, Minnesota
  - Sanofi-Aventis Investigational Site Number 840079, Tupelo, Mississippi
  - Sanofi-Aventis Investigational Site Number 840088, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840060, Syracuse, New York
  - Sanofi-Aventis Investigational Site Number 840029, Charlotte, North Carolina
  - Sanofi-Aventis Investigational Site Number 840074, Bismarck, North Dakota
  - Sanofi-Aventis Investigational Site Number 840026, Cincinnati, Ohio
  - Sanofi-Aventis Investigational Site Number 840078, Dayton, Ohio
  - Sanofi-Aventis Investigational Site Number 840066, Tulsa, Oklahoma
  - Sanofi-Aventis Investigational Site Number 840024, Portland, Oregon
  - Sanofi-Aventis Investigational Site Number 840073, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840022, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840068, Greenville, South Carolina
  - Sanofi-Aventis Investigational Site Number 840071, Cordova, Tennessee
  - Sanofi-Aventis Investigational Site Number 840036, Nashville, Tennessee
  - Sanofi-Aventis Investigational Site Number 840007, San Antonio, Texas
  - Sanofi-Aventis Investigational Site Number 840006, Bennington, Vermont
  - Sanofi-Aventis Investigational Site Number 840089, Seattle, Washington
  - Sanofi-Aventis Investigational Site Number 840020, Charleston, West Virginia
- Australia (7):
  - Sanofi-Aventis Investigational Site Number 036005, Bedford Park
  - Sanofi-Aventis Investigational Site Number 036006, Chatswood
  - Sanofi-Aventis Investigational Site Number 036003, Fitzroy
  - Sanofi-Aventis Investigational Site Number 036004, Geelong
  - Sanofi-Aventis Investigational Site Number 036008, Heidelberg
  - Sanofi-Aventis Investigational Site Number 036002, New Lambton
  - Sanofi-Aventis Investigational Site Number 036001, Sydney
- Sanofi-Aventis Investigational Site Number 040001, Vienna, Austria
- Belarus (5):
  - Sanofi-Aventis Investigational Site Number 112105, Grodno
  - Sanofi-Aventis Investigational Site Number 112102, Minsk
  - Sanofi-Aventis Investigational Site Number 112101, Minsk
  - Sanofi-Aventis Investigational Site Number 112104, Minsk
  - Sanofi-Aventis Investigational Site Number 112103, Vitebsk
- Belgium (4):
  - Sanofi-Aventis Investigational Site Number 056004, Bruges
  - Sanofi-Aventis Investigational Site Number 056002, Leuven
  - Sanofi-Aventis Investigational Site Number 056001, Melsbroek
  - Sanofi-Aventis Investigational Site Number 056003, Sijsele-Damme
- Canada (7):
  - Sanofi-Aventis Investigational Site Number 124004, Gatineau
  - Sanofi-Aventis Investigational Site Number 124002, Kingston
  - Sanofi-Aventis Investigational Site Number 124007, Montreal
  - Sanofi-Aventis Investigational Site Number 124008, Ottawa
  - Sanofi-Aventis Investigational Site Number 124001, Québec
  - Sanofi-Aventis Investigational Site Number 124003, Regina
  - Sanofi-Aventis Investigational Site Number 124006, Saint John
- Chile (3):
  - Sanofi-Aventis Investigational Site Number 152006, Santiago
  - Sanofi-Aventis Investigational Site Number 152007, Santiago
  - Sanofi-Aventis Investigational Site Number 152002, Viña del Mar
- China (32):
  - Sanofi-Aventis Investigational Site Number 156023, Baotou
  - Sanofi-Aventis Investigational Site Number 156031, Beijing
  - Sanofi-Aventis Investigational Site Number 156006, Beijing
  - Sanofi-Aventis Investigational Site Number 156010, Beijing
  - Sanofi-Aventis Investigational Site Number 156005, Beijing
  - Sanofi-Aventis Investigational Site Number 156032, Beijing
  - Sanofi-Aventis Investigational Site Number 156024, Beijing
  - Sanofi-Aventis Investigational Site Number 156030, Beijing
  - Sanofi-Aventis Investigational Site Number 156001, Beijing
  - Sanofi-Aventis Investigational Site Number 156008, Beijing
  - Sanofi-Aventis Investigational Site Number 156007, Changchun
  - Sanofi-Aventis Investigational Site Number 156002, Chengdu
  - Sanofi-Aventis Investigational Site Number 156025, Guangzhou
  - Sanofi-Aventis Investigational Site Number 156012, Guangzhou
  - Sanofi-Aventis Investigational Site Number 156027, Haikou
  - Sanofi-Aventis Investigational Site Number 156021, Hangzhou
  - Sanofi-Aventis Investigational Site Number 156033, Jinan
  - Sanofi-Aventis Investigational Site Number 156034, Nanjing
  - Sanofi-Aventis Investigational Site Number 156011, Nanjing
  - Sanofi-Aventis Investigational Site Number 156019, Qingdao
  - Sanofi-Aventis Investigational Site Number 156029, Shanghai
  - Sanofi-Aventis Investigational Site Number 156016, Shanghai
  - Sanofi-Aventis Investigational Site Number 156009, Shenyang
  - Sanofi-Aventis Investigational Site Number 156022, Shijiazhuang
  - Sanofi-Aventis Investigational Site Number 156018, Suzhou
  - Sanofi-Aventis Investigational Site Number 156028, Taiyuan
  - Sanofi-Aventis Investigational Site Number 156003, Tianjin
  - Sanofi-Aventis Investigational Site Number 156035, Tianjin
  - Sanofi-Aventis Investigational Site Number 156017, Wenzhou
  - Sanofi-Aventis Investigational Site Number 156004, Wuhan
  - Sanofi-Aventis Investigational Site Number 156014, Xi'an
  - Sanofi-Aventis Investigational Site Number 156015, Xi'an
- Czechia (3):
  - Sanofi-Aventis Investigational Site Number 203001, Brno
  - Sanofi-Aventis Investigational Site Number 203002, Ostrava - Poruba
  - Sanofi-Aventis Investigational Site Number 203004, Teplice
- Estonia (2):
  - Sanofi-Aventis Investigational Site Number 233002, Tallinn
  - Sanofi-Aventis Investigational Site Number 233001, Tartu
- France (7):
  - Sanofi-Aventis Investigational Site Number 250005, Besançon
  - Sanofi-Aventis Investigational Site Number 250008, Dijon
  - Sanofi-Aventis Investigational Site Number 250001, Lyon
  - Sanofi-Aventis Investigational Site Number 250007, Nantes
  - Sanofi-Aventis Investigational Site Number 250006, Nice
  - Sanofi-Aventis Investigational Site Number 250002, Nîmes
  - Sanofi-Aventis Investigational Site Number 250003, Poissy
- Germany (9):
  - Sanofi-Aventis Investigational Site Number 276010, Bamberg
  - Sanofi-Aventis Investigational Site Number 276003, Bayreuth
  - Sanofi-Aventis Investigational Site Number 276005, Berlin
  - Sanofi-Aventis Investigational Site Number 276001, Erlangen
  - Sanofi-Aventis Investigational Site Number 276006, Giessen
  - Sanofi-Aventis Investigational Site Number 276004, Hanover
  - Sanofi-Aventis Investigational Site Number 276007, Leipzig
  - Sanofi-Aventis Investigational Site Number 276009, Magdeburg
  - Sanofi-Aventis Investigational Site Number 276002, Wiesbaden
- Greece (2):
  - Sanofi-Aventis Investigational Site Number 300001, Athens
  - Sanofi-Aventis Investigational Site Number 300006, Thessaloniki
- Mexico (2):
  - Sanofi-Aventis Investigational Site Number 484003, México
  - Sanofi-Aventis Investigational Site Number 484005, Monterrey
- Netherlands (5):
  - Sanofi-Aventis Investigational Site Number 528003, 's-Hertogenbosch
  - Sanofi-Aventis Investigational Site Number 528001, Breda
  - Sanofi-Aventis Investigational Site Number 528002, Groesbeek
  - Sanofi-Aventis Investigational Site Number 528004, Nieuwegein
  - Sanofi-Aventis Investigational Site Number 528006, Sittard-Geleen
- Philippines (4):
  - Sanofi-Aventis Investigational Site Number 608004, Cebu City
  - Sanofi-Aventis Investigational Site Number 608002, Makati City
  - Sanofi-Aventis Investigational Site Number 608001, Manila
  - Sanofi-Aventis Investigational Site Number 608003, Quezon City
- Poland (5):
  - Sanofi-Aventis Investigational Site Number 616002, Gdansk
  - Sanofi-Aventis Investigational Site Number 616005, Lodz
  - Sanofi-Aventis Investigational Site Number 616001, Lublin
  - Sanofi-Aventis Investigational Site Number 616004, Szczecin
  - Sanofi-Aventis Investigational Site Number 616003, Warsaw
- Romania (4):
  - Sanofi-Aventis Investigational Site Number 642006, Bacau
  - Sanofi-Aventis Investigational Site Number 642005, Brasov
  - Sanofi-Aventis Investigational Site Number 642001, Bucharest
  - Sanofi-Aventis Investigational Site Number 642007, Oradea
- Slovakia (4):
  - Sanofi-Aventis Investigational Site Number 703003, Bratislava
  - Sanofi-Aventis Investigational Site Number 703005, Bratislava
  - Sanofi-Aventis Investigational Site Number 703001, Martin
  - Sanofi-Aventis Investigational Site Number 703006, Prešov
- Spain (5):
  - Sanofi-Aventis Investigational Site Number 724001, Barcelona
  - Sanofi-Aventis Investigational Site Number 724007, Getafe
  - Sanofi-Aventis Investigational Site Number 724002, Girona
  - Sanofi-Aventis Investigational Site Number 724004, Madrid
  - Sanofi-Aventis Investigational Site Number 724003, Seville
- Sweden (3):
  - Sanofi-Aventis Investigational Site Number 752002, Stockholm
  - Sanofi-Aventis Investigational Site Number 752001, Stockholm
  - Sanofi-Aventis Investigational Site Number 752003, Stockholm
- Thailand (2):
  - Sanofi-Aventis Investigational Site Number 764001, Bangkok
  - Sanofi-Aventis Investigational Site Number 764002, Bangkok Noi
- Tunisia (4):
  - Sanofi-Aventis Investigational Site Number 788003, Manouba
  - Sanofi-Aventis Investigational Site Number 788004, Sfax
  - Sanofi-Aventis Investigational Site Number 788002, Tunis
  - Sanofi-Aventis Investigational Site Number 788001, Tunis
- Turkey (Türkiye) (10):
  - Sanofi-Aventis Investigational Site Number 792011, Edirne
  - Sanofi-Aventis Investigational Site Number 792009, Istanbul
  - Sanofi-Aventis Investigational Site Number 792001, Istanbul
  - Sanofi-Aventis Investigational Site Number 792007, Istanbul
  - Sanofi-Aventis Investigational Site Number 792010, Istanbul
  - Sanofi-Aventis Investigational Site Number 792012, Izmir
  - Sanofi-Aventis Investigational Site Number 792002, Kocaeli
  - Sanofi-Aventis Investigational Site Number 792003, Manisa
  - Sanofi-Aventis Investigational Site Number 792005, Samsun
  - Sanofi-Aventis Investigational Site Number 792004, Trabzon
- Ukraine (19):
  - Sanofi-Aventis Investigational Site Number 804101, Chernihiv
  - Sanofi-Aventis Investigational Site Number 804103, Dnipropetrovsk
  - Sanofi-Aventis Investigational Site Number 804107, Donetsk
  - Sanofi-Aventis Investigational Site Number 804117, Donetsk
  - Sanofi-Aventis Investigational Site Number 804119, Ivano-Frankivsk
  - Sanofi-Aventis Investigational Site Number 804102, Kharkiv
  - Sanofi-Aventis Investigational Site Number 804109, Kharkiv
  - Sanofi-Aventis Investigational Site Number 804115, Kiev
  - Sanofi-Aventis Investigational Site Number 804116, Kiev
  - Sanofi-Aventis Investigational Site Number 804108, Kiev
  - Sanofi-Aventis Investigational Site Number 804111, Lutsk
  - Sanofi-Aventis Investigational Site Number 804124, Lutsk
  - Sanofi-Aventis Investigational Site Number 804114, Lviv
  - Sanofi-Aventis Investigational Site Number 804121, Lviv
  - Sanofi-Aventis Investigational Site Number 804120, Poltava
  - Sanofi-Aventis Investigational Site Number 804105, Vinnytsia
  - Sanofi-Aventis Investigational Site Number 804118, Zaporizhya
  - Sanofi-Aventis Investigational Site Number 804104, Zaporizhzhia
  - Sanofi-Aventis Investigational Site Number 804122, Zaporizhzhya
- United Kingdom (5):
  - Sanofi-Aventis Investigational Site Number 826002, Edinburgh
  - Sanofi-Aventis Investigational Site Number 826004, Haywards Heath
  - Sanofi-Aventis Investigational Site Number 826001, Irvine
  - Sanofi-Aventis Investigational Site Number 826003, Leeds
  - Sanofi-Aventis Investigational Site Number 826005, Salford

REFERENCES:
- [Result] Confavreux C, O'Connor P, Comi G, Freedman MS, Miller AE, Olsson TP, Wolinsky JS, Bagulho T, Delhay JL, Dukovic D, Truffinet P, Kappos L; TOWER Trial Group. Oral teriflunomide for patients with relapsing multiple sclerosis (TOWER): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2014 Mar;13(3):247-56. doi: 10.1016/S1474-4422(13)70308-9. Epub 2014 Jan 23. PMID 24461574
- [Derived] Comi G, Freedman MS, Meca-Lallana JE, Vermersch P, Kim BJ, Parajeles A, Edwards KR, Gold R, Korideck H, Chavin J, Poole EM, Coyle PK. Prior treatment status: impact on the efficacy and safety of teriflunomide in multiple sclerosis. BMC Neurol. 2020 Oct 6;20(1):364. doi: 10.1186/s12883-020-01937-4. PMID 33023488
- [Derived] Miller AE, Olsson TP, Wolinsky JS, Comi G, Kappos L, Hu X, Xu X, Lublin AL, Truffinet P, Chavin J, Delhay JL, Benamor M, Purvis A, Freedman MS; TOWER investigators. Long-term safety and efficacy of teriflunomide in patients with relapsing multiple sclerosis: Results from the TOWER extension study. Mult Scler Relat Disord. 2020 Nov;46:102438. doi: 10.1016/j.msard.2020.102438. Epub 2020 Aug 1. PMID 32911306
- [Derived] Qiu W, Huang DH, Hou SF, Zhang MN, Jin T, Dong HQ, Peng H, Zhang CD, Zhao G, Huang YN, Zhou D, Wu WP, Wang BJ, Li JM, Zhang XH, Cheng Y, Li HF, Li L, Lu CZ, Zhang X, Bu BT, Dong WL, Fan DS, Hu XQ, Xu XH; TOWER Trial Chinese Group. Efficacy and Safety of Teriflunomide in Chinese Patients with Relapsing Forms of Multiple Sclerosis: A Subgroup Analysis of the Phase 3 TOWER Study. Chin Med J (Engl). 2018 Dec 5;131(23):2776-2784. doi: 10.4103/0366-6999.246067. PMID 30511679
- [Derived] Freedman MS, Morawski J, Thangavelu K. Clinical efficacy of teriflunomide over a fixed 2-year duration in the TOWER study. Mult Scler J Exp Transl Clin. 2018 May 16;4(2):2055217318775236. doi: 10.1177/2055217318775236. eCollection 2018 Apr-Jun. PMID 29796289
- [Derived] Freedman MS, Wolinsky JS, Comi G, Kappos L, Olsson TP, Miller AE, Thangavelu K, Benamor M, Truffinet P, O'Connor PW; TEMSO and TOWER Study Groups. The efficacy of teriflunomide in patients who received prior disease-modifying treatments: Subgroup analyses of the teriflunomide phase 3 TEMSO and TOWER studies. Mult Scler. 2018 Apr;24(4):535-539. doi: 10.1177/1352458517695468. Epub 2017 Mar 17. PMID 28304217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1493 participants were screened at 193 sites in 26 countries. The common end date for core treatment period was on 17 April 2012 (maximum treatment duration of 173 weeks). The extension study was completed on 18 June 2015 (maximum treatment duration was 174 weeks in addition to core treatment period).
Pre-assignment Details: Randomization was stratified by investigational site and Expanded Disability Status Scale (EDSS) score ≤3.5 or >3.5). Assignment to groups was done using an Interactive Voice Response System(IVRS) in 1:1:1 ratio. 1169 participants were randomized at 190 sites. 780 participants completed core treatment period and 751 were treated in extension study.
Period: Core Treatment Period
Arm/Group | Placebo / Teriflunomide 14 mg | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg
Started | 389 (Randomized) | 408 (Randomized) | 372 (Randomized)
Treated | 388 (1 participant received teriflunomide 7 mg and 2 participants teriflunomide 14 mg (at least 1 dose)) | 407 (1 participant received placebo (at least 1 dose)) | 370 (1 participant received teriflunomide 7 mg and 1 participant placebo (at least 1 dose))
Completed | 263 | 273 | 244
Not Completed | 126 | 135 | 128
Not completed — Not treated | 1 | 1 | 2
Not completed — Adverse Event | 26 | 54 | 58
Not completed — Lack of Efficacy | 37 | 30 | 20
Not completed — Poor compliance to protocol | 15 | 3 | 4
Not completed — Lost to Follow-up | 6 | 4 | 3
Not completed — Other: protocol deviation | 3 | 3 | 7
Not completed — Other: wish to parent | 5 | 7 | 4
Not completed — Other: personal/family constraints | 6 | 7 | 10
Not completed — Other: MS treatment change | 6 | 4 | 4
Not completed — Other: tolerability complaints | 2 | 0 | 0
Not completed — Other:participant's decision/unspecified | 19 | 22 | 16
Period: Extension Study Period
Arm/Group | Placebo / Teriflunomide 14 mg | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg
Started | 253 (10 participants completed core treatment period but did not enter in extension treatment period.) | 265 (8 participants completed core treatment period but did not enter in extension treatment period.) | 233 (11 participants completed core treatment period but did not enter in extension treatment period.)
Completed | 188 | 194 | 167
Not Completed | 65 | 71 | 66
Not completed — Adverse Event | 18 | 20 | 21
Not completed — Lack of Efficacy | 14 | 10 | 20
Not completed — Lost to Follow-up | 4 | 9 | 6
Not completed — Poor Compliance to Protocol | 3 | 2 | 1
Not completed — Other than specified above | 26 | 30 | 18

BASELINE CHARACTERISTICS:
Groups:
- Placebo / Teriflunomide 14 mg: Core treatment period: Placebo once daily. Extension treatment period: Teriflunomide 14 mg once daily.
- Total: Total of all reporting groups
Arm/Group | Placebo / Teriflunomide 14 mg | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg | Total
Number analyzed (Participants) | 389 | 408 | 372 | 1169
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (9.1) | 37.4 (9.4) | 38.2 (9.4) | 37.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273 | 300 | 258 | 831
  Male | 116 | 108 | 114 | 338
Region of Enrollment [Number; unit: participants] — Due to the small sample size in some countries, the countries were pooled as follows:
  * Eastern Europe: Belarus, Czech Republic, Estonia, Greece, Poland, Romania, Slovakia and Ukraine
  * Western Europe and Africa: Austria, Belgium, France, Germany, Netherlands, Spain, Sweden and United Kingdom, Tunisia and Turkey
  * Asia and Australia: China, Philippines, Thailand and Australia
  * America: Canada, Chile, Mexico and the USA
  participants
    Eastern Europe | 117 | 124 | 116 | 357
    Western Europe and Africa | 121 | 127 | 120 | 368
    Asia and Australia | 67 | 65 | 55 | 187
    America | 84 | 92 | 81 | 257
Time since first diagnosis of Multiple Sclerosis (MS) [Mean (Standard Deviation); unit: years] — The information was not available for one participant in the teriflunomide 14 mg group
  years | 4.92 (5.66) | 5.30 (5.45) | 5.27 (5.90) | 5.16 (5.66)
Number of MS relapses [Median (Full Range); unit: relapses] — The information was not available for:
  * 'Within the past year': 1 participant in the placebo group and 1 participant in the teriflunomide 14 mg group
  * 'Within the past 2 years': 2 participants in the teriflunomide 14 mg group
  relapses
    Within the past year | 1 [0 to 7] | 1 [0 to 5] | 1 [0 to 5] | 1 [0 to 7]
    Within the past 2 years | 2 [1 to 8] | 2 [1 to 8] | 2 [1 to 9] | 2 [1 to 9]
Time since most recent MS relapse onset [Mean (Standard Deviation); unit: months] — The information was not available for one participant in the teriflunomide 14 mg group.
  months | 5.29 (3.41) | 5.18 (3.41) | 5.33 (3.32) | 5.26 (3.38)
MS subtype [Number; unit: participants]
  Relapsing Remitting | 379 | 393 | 366 | 1138
  Secondary Progressive | 4 | 3 | 2 | 9
  Progressive Relapsing | 6 | 12 | 2 | 20
  Information not available | 0 | 0 | 2 | 2
Baseline EDSS score [Number; unit: participants] — EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation.
  EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  participants
    ≤3.5 | 294 | 301 | 276 | 871
    >3.5 | 95 | 107 | 96 | 298

OUTCOME MEASURES:

1. Primary Outcome: Core Treatment Period: Annualized Relapse Rate (ARR): Poisson Regression Estimate
Description: ARR is obtained from the total number of confirmed relapses that occurred during the treatment period divided by the sum of treatment durations.
  Each episode of relapse - appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever - was to be confirmed by an increase in Expanded Disability Status Scale (EDSS) score or Functional System scores.
  To account for the different treatment durations among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses as response variable; log-transformed treatment duration as "offset" variable; treatment group, region of enrollment and baseline EDSS stratum as covariates).
Time Frame: Core treatment period between 48 - 152 weeks depending on time of enrollment
Population: Intent-to-treat population: all randomized and treated participants. Participants were considered in the treatment group to which they were randomized regardless of the drug they actually received.
Measure: Number (95% Confidence Interval); unit: relapses per year
Groups:
- Placebo: Placebo once daily
- Teriflunomide 7 mg: Teriflunomide 7 mg once daily
- Teriflunomide 14 mg: Teriflunomide 14 mg once daily
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
relapses per year | 0.501 [0.432 to 0.581] | 0.389 [0.332 to 0.457] | 0.319 [0.267 to 0.381]
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; Null hypothesis: * H1: No difference between teriflunomide 14 mg and placebo * H2: No difference between teriflunomide 7 mg and placebo The study was sized to have 94% power to detect a 25% relative risk reduction in ARR with teriflunomide compared to placebo at a 2-sided 0.05 significance level; Test type: Superiority or Other; p = 0.0001, Regression, Poisson — Step down approach used to adjust for multiplicity: * H1 tested first * H2 tested only if the comparison H1 was statistically significant A priori threshold for statistical significance for both comparisons ≤0.05; Relative risk reduction (%) = 36.3 — Relative risk reduction with teriflunomide 14 mg compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; Test type: Superiority or Other; p = 0.0183, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; Relative Risk Reduction (%) = 22.3 — Relative risk reduction with teriflunomide 7 mg compared to placebo

2. Secondary Outcome: Core Treatment Period: Time to Disability Progression
Description: Probability of disability progression at 24, 48, 108 and 132 weeks was estimated using Kaplan-Meier method on the time to disability progression defined as the time from randomization to first 12-week sustained disability progression [i.e. increase from baseline of at least 1 point in EDSS score (at least 0.5 point for participants with baseline EDSS score >5.5) that persisted for at least 12 weeks].
  Participants free of disability progression (no disability progression observed on treatment) were censored at the date of the last on-treatment EDSS evaluation.
  Kaplan-Meier method consists in computing probabilities of non occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time t. Probability of event at time t is 1 minus the probability of being event-free for the amount of time t.
Time Frame: Core treatment period between 48 - 152 weeks depending on time of enrollment
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
percent probability
  Probability of disability progression at 24 weeks | 8.0 [5.2 to 10.7] | 5.3 [3.0 to 7.6] | 2.7 [0.9 to 4.4]
  Probability of disability progression at 48 weeks | 14.2 [10.6 to 17.9] | 12.1 [8.7 to 15.5] | 7.8 [4.9 to 10.8]
  Probability of disability progression at 108 weeks | 19.7 [15.2 to 24.1] | 21.1 [16.1 to 26.1] | 15.8 [11.2 to 20.4]
  Probability of disability progression at 132 weeks | 21.0 [15.9 to 26.0] | 22.2 [16.8 to 27.6] | 15.8 [11.2 to 20.4]
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; Null hypothesis: * S1: No difference between teriflunomide 14 mg and placebo * S2: No difference between teriflunomide 7 mg and placebo The study was also sized to have 75% power to detect a 37% hazard ratio reduction in time to disability progression with teriflunomide compared to placebo; Test type: Superiority or Other; p = 0.0442, Log Rank — Step down approach: * S1 tested only if both comparisons on the primary outcome measure were statistically significant * S2 tested only if the comparison S1 was statistically significant A priori threshold for statistical significance ≤0.05; Two-sided Log-rank test stratified by region of enrollment and baseline EDSS stratum; Hazard ratio reduction (%) = 31.5 — Relative reduction in the hazard rate with teriflunomide 14 mg compared to placebo (estimated from a Cox proportional hazard model with treatment arm, region of enrollment and baseline EDSS stratum as covariates)
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; Test type: Superiority or Other; p = 0.7620, Log Rank — [p-value comment as in outcome 2, analysis 1]; Two-sided Log-rank test stratified by region of enrollment and baseline EDSS stratum; Hazard ratio reduction (%) = 4.5 — Relative reduction in the hazard rate with teriflunomide 7 mg compared to placebo (estimated from a Cox proportional hazard model with treatment arm, region of enrollment and baseline EDSS stratum as covariates)

3. Secondary Outcome: Core Treatment Period: Time Without Relapse
Description: Probability of no relapse at 24, 48, 108 and 132 weeks was estimated using Kaplan-Meier method on the time to relapse defined as the time from randomization to first EDSS confirmed relapse.
  Participants free of confirmed relapse (no EDSS confirmed relapse observed on treatment) were censored at the date of the last study drug intake.
Time Frame: Core treatment period between 48 - 152 weeks depending on time of enrollment
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
percent probability
  Probability of no relapse at 24 weeks | 76.4 [72.1 to 80.7] | 81.5 [77.6 to 85.4] | 85.5 [81.8 to 89.2]
  Probability of no relapse at 48 weeks | 60.6 [55.5 to 65.6] | 71.9 [67.3 to 76.5] | 76.3 [71.7 to 81.0]
  Probability of no relapse at 108 weeks | 46.8 [41.0 to 52.6] | 58.2 [52.6 to 63.8] | 57.1 [50.5 to 63.7]
  Probability of no relapse at 132 weeks | 37.7 [30.2 to 45.2] | 55.4 [48.8 to 62.0] | 51.5 [43.6 to 59.5]

4. Secondary Outcome: Core Treatment Period: Change From Baseline to Week 48 in EDSS Total Score
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation.
  EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  Baseline adjusted least-squares means at Week 48 were estimated using a Mixed-effect model with repeated measures (MMRM) on EDSS score data (treatment group, region of enrollment, baseline EDSS stratum, visit, treatment-by-visit interaction, baseline value, and baseline-by-visit interaction as factors). All the timepoints from randomization up to Week 48 were included in the model.
Time Frame: Baseline (before randomization), Week 12, Week 24, Week 36 and Week 48
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
units on a scale | 0.089 (0.050) | 0.042 (0.049) | -0.050 (0.052)

5. Secondary Outcome: Core Treatment Period: Change From Baseline to Week 48 in Fatigue Impact Scale (FIS) Total Score
Description: FIS is a participants-reported scale that qualifies the impact of fatigue on daily life in participants with MS. It consists of 40 statements that measure fatigue in 3 areas; physical, cognitive, and social.
  FIS total score ranges from 0 (no problem) to 160 (extreme problem).
  Baseline adjusted least-squares means at week 48 were estimated using a Mixed-effect model with repeated measures (MMRM) on FIS total score data (treatment group, region of enrollment, baseline EDSS stratum, visit, treatment-by-visit interaction, baseline value, and baseline-by-visit interaction as factors). All the timepoints from randomization up to Week 48 were included in the model.
Time Frame: Baseline (before randomization), Week 12, Week 24 and Week 48
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
units on a scale | 4.669 (1.576) | 2.512 (1.533) | 1.915 (1.628)

6. Secondary Outcome: Core Treatment Period: Change From Baseline to Last Visit in Fatigue Impact Scale (FIS) Total Score
Description: Baseline adjusted least-squares means at last visit were estimated using an analysis of covariance (ANCOVA) model on collected data for FIS total score (treatment group, region of enrollment, baseline EDSS stratum, visit number for the last visit and baseline value as factors).
Time Frame: Baseline (before randomization) and up to Week 152
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
units on a scale | 6.311 (1.671) | 4.464 (1.657) | 2.043 (1.682)

7. Secondary Outcome: Core Treatment Period: Change From Baseline to Week 48 in Short Form Generic Health Survey - 36 Items (SF-36) Summary Scores
Description: SF-36 scale is a generic, self-administered, health-related quality-of-life (QOL) instrument. It is constructed such that the 36 questions represent 8 of the most important health concepts: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
  Two summary scores are obtained:
  * the physical health component summary score,
  * the mental health component summary score.
  Both scores range from 0 to 100 and a high score indicates a more favorable health state.
  Baseline adjusted least-squares means at week 48 were estimated using a Mixed-effect model with repeated measures [MMRM] on each summary score data (treatment group, region of enrollment, baseline EDSS stratum, visit, treatment-by-visit interaction, baseline value, and baseline-by-visit interaction as factors). All the timepoints from randomization up to Week 48 were included in the model.
Time Frame: Baseline (before randomization), Week 12, Week 24 and Week 48
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
units on a scale
  Physical health component | -1.082 (0.405) | -0.397 (0.396) | -0.105 (0.418)
  Mental health component | -2.913 (0.586) | -2.031 (0.571) | -1.434 (0.606)

8. Secondary Outcome: Core Treatment Period: Change From Baseline to Last Visit in Short Form Generic Health Survey - 36 Items (SF-36) Summary Scores
Description: Baseline adjusted least-squares means at last visit were estimated using an analysis of covariance (ANCOVA) model on collected data for each summary score (treatment group, region of enrollment, baseline EDSS stratum, visit number for the last visit and baseline value as factors).
Time Frame: Baseline (before randomization) and up to Week 152
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 388 | 407 | 370
units on a scale
  Physical Health component | -1.629 (0.435) | -0.909 (0.441) | -0.638 (0.436)
  Mental Health component | -2.792 (0.592) | -1.704 (0.597) | -1.087 (0.593)

9. Secondary Outcome: Core Treatment Period: Overview of Adverse Events
Description: Adverse Events (AE) are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: From first study drug intake up to 112 days after last intake in the core treatment period or up to first intake in the extension treatment period, whichever occurred first
Population: All randomized and treated participants. Participants were considered according to the drug actually received.
  The 3 participants in the placebo group who received teriflunomide were analyzed according to the teriflunomide dose.
  The participant in the teriflunomide 14 mg group who received 7 mg was analyzed in the teriflunomide 7 mg group.
Measure: Number; unit: participants
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 385 | 409 | 371
participants
  Any AE | 320 | 344 | 320
  - Any serious AE | 47 | 52 | 44
  - Any AE leading to death | 1 | 1 | 2
  - Any AE leading to treatment discontinuation | 24 | 53 | 58

10. Secondary Outcome: Extension Treatment Period: Overview of Treatment Emergent Adverse Events (TEAE)
Description: AEs were any unfavourable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: From first intake of study drug in extension treatment period up to 28 days after the last intake in the extension treatment period
Population: Safety population: all randomized participants who received at least 1 dose of investigational product.
  Two participants in placebo of core study received teriflunomide and were analyzed according to teriflunomide dose.
  One participant in teriflunomide 14 mg in core study group who received 7 mg was analyzed in teriflunomide 7 mg group.
Measure: Number; unit: participants
Arm/Group | Placebo / Teriflunomide 14 mg | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg
Number analyzed (Participants) | 251 | 267 | 233
participants
  Any TEAE | 203 | 200 | 188
  Any serious TEAE | 16 | 33 | 29
  Any TEAE leading to death | 1 | 3 | 1
  Any TEAE leading to treatment discontinuation | 17 | 17 | 20

11. Secondary Outcome: Extension Treatment Period: Time to Disability Progression
Description: Probability of disability progression since the randomization of the core period was estimated using Kaplan-Meier method on the time to disability progression defined as the time from randomization to first 12 week sustained disability progression [i.e. increase from baseline of at least 1 point in EDSS score (at least 0.5 point for participants with baseline EDSS score >5.5) that persisted for at least 12 weeks].
  Participants free of disability progression (no disability progression observed on treatment) were censored at the date of the last on-treatment EDSS evaluation.
  Kaplan-Meier method consists in computing probabilities of non occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event free for the amount of time t. Probability of event at time t was 1 minus the probability of being event-free for the amount of time t.
Time Frame: Core treatment period (maximum: 173 weeks) and Extension treatment period (maximum: 174 weeks)
Population: ITT population for extension treatment period consists of all participants with a signed informed consent form for the extension and with a date of treatment allocated or recorded in the IVRS/IWRS database, regardless of whether the treatment was actually taken.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo / Teriflunomide 14 mg | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg
Number analyzed (Participants) | 253 | 265 | 233
percent probability
  1 year | 0.130 [0.089 to 0.172] | 0.117 [0.078 to 0.156] | 0.077 [0.043 to 0.112]
  2 year | 0.190 [0.142 to 0.238] | 0.175 [0.129 to 0.221] | 0.147 [0.101 to 0.192]
  3 year | 0.245 [0.191 to 0.299] | 0.233 [0.181 to 0.285] | 0.190 [0.139 to 0.241]
  4 year | 0.307 [0.246 to 0.368] | 0.270 [0.214 to 0.326] | 0.248 [0.189 to 0.307]
  5 year | 0.328 [0.262 to 0.395] | 0.317 [0.250 to 0.384] | 0.265 [0.203 to 0.327]

12. Secondary Outcome: Extension Treatment Period: ARR: Poisson Regression Estimate
Description: ARR was obtained from the total number of confirmed relapses that occurred during the treatment period divided by the sum of treatment durations. A relapse is defined as the appearance of a new clinical sign/symptom or clinical worsening of a previous sign/symptom (one that had been stable for at least 30 days) that persists for a minimum of 24 hours in the absence of fever. Relapse was confirmed by an increase in EDSS score or Functional System scores. To account for the different treatment durations among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses as response variable; log-transformed treatment duration as "offset" variable; treatment group, region of enrolment and baseline EDSS stratum as covariates).
Time Frame: Extension treatment period (Maximum: 174 weeks)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Placebo / Teriflunomide 14 mg | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg
Number analyzed (Participants) | 253 | 265 | 233
relapses per year | 0.199 [0.156 to 0.254] | 0.200 [0.155 to 0.257] | 0.179 [0.132 to 0.243]

13. Other Pre Specified Outcome: Core Treatment Period: Liver Function: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA)
Description: PCSA values are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review.
  Hepatic parameters thresholds were defined as follows:
  * Alanine Aminotransferase (ALT) >3, 5, 10 or 20 upper limit of normal(ULN);
  * Aspartate aminotransferase (AST) >3, 5, 10 or 20 ULN;
  * Alkaline Phosphatase >1.5 ULN;
  * Total Bilirubin (TB) >1.5 or 2 ULN;
  * ALT >3 ULN and TB >2 ULN.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 385 | 409 | 371
participants
  ALT >3 ULN | 22 | 31 | 29
  - ALT >5 ULN | 14 | 10 | 11
  - ALT >10 ULN | 5 | 2 | 3
  AST >3 ULN | 13 | 9 | 9
  - AST >5 ULN | 9 | 3 | 3
  Alkaline Phosphatase >1.5 ULN | 5 | 4 | 2
  TB >1.5 ULN | 9 | 6 | 8
  ALT >3 ULN and TB >2 ULN | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from signature of the Informed Consent Form up to the last visit (174 weeks) in the study.
Description: The analysis was performed on the safety population as previously defined and included all AE that developed or worsened and death that occurred during first intake of study drug in extension treatment period up to 28 days after the last intake in the extension study treatment period.
Groups:
- Placebo / 14 mg: Core treatment period: Placebo once daily. Extension treatment period: Teriflunomide 14 mg once daily
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg | Placebo / 14 mg | Teriflunomide 7 mg / 14 mg | Teriflunomide 14 mg / 14 mg
Serious Adverse Events (participants affected / at risk) | 47/385 | 52/409 | 44/371 | 16/251 | 33/267 | 29/233
Other Adverse Events (participants affected / at risk) | 247/385 | 270/409 | 254/371 | 152/251 | 153/267 | 138/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=385) | Teriflunomide 7 mg (N=409) | Teriflunomide 14 mg (N=371) | Placebo / 14 mg (N=251) | Teriflunomide 7 mg / 14 mg (N=267) | Teriflunomide 14 mg / 14 mg (N=233)
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Abscess soft tissue (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Endocarditis enterococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infected bites (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Neuroborreliosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Perichondritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 2 | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 3 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 2 | 1 | 1 | 1 | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastropleural fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stress ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic dysplasia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Choledochal cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Congenital flat feet (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 6 | 3 | 2 | 1 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=385) | Teriflunomide 7 mg (N=409) | Teriflunomide 14 mg (N=371) | Placebo / 14 mg (N=251) | Teriflunomide 7 mg / 14 mg (N=267) | Teriflunomide 14 mg / 14 mg (N=233)
Nasopharyngitis (Infections and infestations) | 65 | 51 | 44 | 22 | 21 | 22
Influenza (Infections and infestations) | 19 | 22 | 22 | 8 | 14 | 16
Urinary tract infection (Infections and infestations) | 36 | 38 | 26 | 8 | 12 | 10
Sinusitis (Infections and infestations) | 16 | 25 | 24 | 5 | 10 | 9
Upper respiratory tract infection (Infections and infestations) | 42 | 35 | 33 | 11 | 12 | 7
Neutropenia (Blood and lymphatic system disorders) | 10 | 19 | 18 | 2 | 13 | 20
Depression (Psychiatric disorders) | 25 | 28 | 18 | 8 | 15 | 10
Headache (Nervous system disorders) | 41 | 61 | 47 | 10 | 15 | 17
Hypoaesthesia (Nervous system disorders) | 16 | 22 | 23 | 12 | 6 | 8
Dizziness (Nervous system disorders) | 23 | 17 | 25 | 3 | 8 | 4
Paraesthesia (Nervous system disorders) | 23 | 27 | 22 | 12 | 5 | 4
Hypertension (Vascular disorders) | 8 | 17 | 16 | 10 | 13 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 21 | 12 | 5 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 39 | 45 | 35 | 14 | 18 | 20
Nausea (Gastrointestinal disorders) | 27 | 38 | 36 | 14 | 10 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 42 | 50 | 36 | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 28 | 32 | 12 | 13 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 30 | 20 | 7 | 9 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 19 | 25 | 7 | 9 | 9
Fatigue (General disorders) | 40 | 33 | 37 | 9 | 12 | 6
Alanine aminotransferase increased (Investigations) | 27 | 43 | 48 | 27 | 8 | 9
Fall (Injury, poisoning and procedural complications) | 14 | 22 | 23 | 4 | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can present or publish results. The investigator provides the sponsor with a copy of the presentation or publication for review and comment at least 30 days in advance of its submission.

The sponsor can delay the submission for a period not exceeding 90 days to allow for filing a patent application or such other measures as sponsor deems appropriate to establish and preserve its proprietary rights.